CLINICAL TRIAL: NCT01179074
Title: Palliative Stenting With or Without Radiotherapy for Inoperable Oesophageal Carcinoma: a Randomised Trial
Brief Title: Role of Radiotherapy Following Oesophageal Stenting in Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Prof. T.K.Chattopadhyay, Department of G.I.Surgery, All India Institute of Medical Sciences, New Delhi-110029
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SEMSRT-1
Record Dates: First submitted 2010-05-25; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-02

CONDITIONS: Oesophageal Cancer
Keywords: palliation inoperable oesophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oesophageal stent alone (Active Comparator): Patients of inoperable oesophageal cancer in this arm underwent oesophageal stenting with self expandable metal stents
  Interventions: Procedure: oesophageal stenting with self expandable metal stent
- Oesophageal stent followed by EBRT (Active Comparator): Patients in this arm underwent oesophageal stenting with self expandable metal stents followed by external beam radiotherapy (30Gy/10#/2weeks)
  Interventions: Procedure: oesophageal stenting with self expandable metal stent; Procedure: Oesophageal stent followed by external beam radiotherapy

INTERVENTIONS:
Procedure: oesophageal stenting with self expandable metal stent — oesophageal stent placement for high grade dysphagia in inoperable oesophageal cancer
  Other Names: Ultraflex stent, Microvasive, Boston Scientific
Procedure: Oesophageal stent followed by external beam radiotherapy — 30 Gy in 10 fractions over 2 weeks administered in the stent followed by EBRT group
  Other Names: External beam radiotherapy
  Arms: Oesophageal stent followed by EBRT

SUMMARY:
To assess the benefits of oesophageal stenting and external beam radiotherapy over oesophageal stenting alone in patients with inoperable oesophageal cancer

DETAILED DESCRIPTION:
A majority of patients with oesophageal cancer present with inoperable disease and require rapid and long lasting palliation of dysphagia.

STUDY AIM: To compare dysphagia relief in patients treated with oesophageal stenting and external beam radiotherapy (EBRT), versus oesophageal stenting alone and to assess overall survival, treatment related complications, and quality of life in the two groups.

PATIENTS AND METHODS: Patients with inoperable oesophageal cancer with high grade dysphagia to be randomised to receive oesophageal stenting alone (Group I), versus a combination of stenting followed by EBRT (Group II). Dysphagia relief, treatment related complications, overall survival, and quality of life to be assessed in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Oesophageal cancer patients with locally advanced unresectable cancer (such as invasion of tracheo-bronchial tree, aorta, pulmonary vascular structures, etc),
* Metastatic disease, and co-morbid conditions precluding major surgical procedure (such as severe cardiopulmonary, hepatic and renal diseases) with grade 3 and 4 dysphagia, were included in the trial.

Exclusion Criteria:

* Patients with carcinoma of the cervical oesophagus and those who had already received prior radiotherapy, chemotherapy, or any other modality of treatment were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Relief of dysphagia | 1 week after intervention
  Relief of dysphagia will be assessed by stratifying the ability to swallow into the following grades.
  Grade 1: Difficulty in swallowing solid food Grade 2: Difficulty in swallowing semisolid food Grade 3: Difficulty in swallowing liquids Grade 4: Difficulty in swallowing even saliva The dysphagia scores will be assessed 1 week after intervention (stenting and radiotherapy)in the two groups
Relief of dysphagia | 3 months following intervention
  Dysphagia grades at 3 months will be assessed in the two groups
Relief of dysphagia | 5 months after intervention
  Dysphagia grades at 5 months will be assessed in the two groups

SECONDARY OUTCOMES:
Survival | From the date of diagnosis till death
  Patients will be followed up at baseline, 1 week after oesophageal stenting, 1 week after completion of radiotherapy and 2 monthly thereafter till their death

CONTACTS AND LOCATIONS:
Overall Officials: Tushar K Chattopadhyay, MS, Study Director — Head, Dept. G.I Surgery, All India Institute of Medical Sciences, New Delhi
Locations (1):
- Departments of Gastrointestinal surgery, Gastroenterology, Radiation Oncology, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Schmid EU, Alberts AS, Greeff F, Terblanche AP, Schoeman L, Burger W, Shiels RA, Friediger D, Van der Hoven A, Falkson G. The value of radiotherapy or chemotherapy after intubation for advanced esophageal carcinoma--a prospective randomized trial. Radiother Oncol. 1993 Jul;28(1):27-30. doi: 10.1016/0167-8140(93)90181-7. PMID 7694321